CLINICAL TRIAL: NCT02679027
Title: New Test for Prediction of Difficult Intubation: Tongue Protrusion Movements
Brief Title: Difficult Intubation and Tongue Protrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Alkin Colak, Associate professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: tongueintubation
Record Dates: First submitted 2016-01-27; First posted 2016-02-10 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Difficult Intubation, Tongue Mobility

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Easy intubation (Active Comparator): Intubation difficulty score <5
  Interventions: Other: Protrude tongue maximally and upward (PTMU); Other: Protrude tongue maximally and downward (PTMD)
- Difficult intubation (Active Comparator): Intubation difficulty score >5
  Interventions: Other: Protrude tongue maximally and upward (PTMU); Other: Protrude tongue maximally and downward (PTMD)

INTERVENTIONS:
Other: Protrude tongue maximally and upward (PTMU) — The horizontal line was passing through the mid points of the distance between subnasale to stomion (upper lip height). Patients were asked to protrude tongue maximally and upward (PTMU).
Other: Protrude tongue maximally and downward (PTMD) — The horizontal line was passing through the mid points of the distance between stomion to mentum (mandible height). Patients were asked to protrude tongue maximally and downward (PTMD).

SUMMARY:
Objectives: The aim of study is to determine the possible usage of tongue movements out of the mouth in the prediction of difficult intubation.

Method: Two hundred twenty three patients undergoing abdominal surgery with general anesthesia between 2014 and 2015 were enrolled in this study. Difficult intubation was evaluated using the intubation difficulty scale (IDS) score. All intubations were performed by anesthesiologist to eliminate the differences among the anesthesiologists' experiences. IDS score were evaluated by anesthesiologists who had no idea about the measurements of the tongue movements and performed laryngeal intubation in all patients.

To define the tongue movements, horizontal lines were used. Horizontal line were passing through the mid points of mandible and upper lip height. Patients were asked to protrude tongue maximally and upward (PTMU), to protrude tongue maximally and downward (PTMD) in anatomical neutral position which was sitting down on a chair.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing abdominal surgery with general anesthesia
* Able to sit

Exclusion Criteria:

* Enable to sit,
* Patients had head or neck surgery,
* Patients with unstable cardiological and respiratory hemodynamic symptoms,
* Dental prosthesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Intubation difficulty scale | 2 days
  Intubation difficulty scale score includes 7 variables for difficult intubation. N1: The number of attempts for intubation (for the first attempt 0 point, for the other attempts 1 point each); N2: The number of anesthesiologist for the laryngoscopies (for the first attempt 0 point, for the other attempts 1 point each); N3: Alternative intubation techniques that are used (if not needed 0 point, change of blade type or using blind nasotracheal intubation 1 point each); N4: 1 point less than Cormack and Lehane Classification for defining glottic exposure; N5: The degree of force of lifting laryngoscopy (normal lifting 0 point, more force needed 1 point); N6: Using external laryngeal pressure 1 point; N7: The view of the vocal cords (abduction position 0 point, adduction position 1 point). A score of 0-4 defines easy intubation and an IDS score ≥5 defines difficult intubation